CLINICAL TRIAL: NCT04553289
Title: Exercise Into Pain in Subacromial Shoulder Pain: a Randomized Controlled Trial
Brief Title: Exercise Into Pain in Subacromial Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University of Malaga (Other); Rotterdam University of Applied Sciences (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Filip Struyf, Professor, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18/34/379 (RCT)
Record Dates: First submitted 2020-08-20; First posted 2020-09-17 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Shoulder Impingement Syndrome
Keywords: shoulder pain; subacromial impingement syndrome; exercise therapy
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercising into pain (Experimental): The participants will train during 12 with progressive loaded exercises, three times per week. There are 9 sessions of supervised physiotherapy treatment, lasting 30 minutes, while the rest of the sessions is conducted as home exercises. There are 4 strengthening exercises, including 2 in closed kinetic chain exercises and 2 executed with the elastic band or with dumbbell/weight. One exercise will be performed with pain ranging between 4 and 7 on a NPRS (Numeric Pain Rating Scale) and the rest of the exercises will be performed with no/slight pain, ranging between 0 and 2 on NPRS. At week 9, patients will continue to exercise with pain between 0 and 2 in all exercises. 10/15 minutes of manual therapy (posterior capsular release) will be applied during the physiotherapy session.
  Interventions: Other: exercising into pain
- exercising with no/slight pain (Active Comparator): The participants will train during 12 weeks with progressive loaded exercises, three times per week. There are 9 sessions of supervised physiotherapy treatment, lasting 30 minutes, while the rest of the sessions is conducted as home exercises. There are 4 strengthening exercises, including 2 in closed kinetic chain exercises and 2 executed with the elastic band or with dumbbell/weight. All the exercises will be performed with no/slight pain, ranging between 0 and 2 on NPRS. 10/15 minutes of manual therapy (posterior capsular release) will be applied during the physiotherapy session.
  Interventions: Other: exercising with no/slight pain

INTERVENTIONS:
Other: exercising into pain — the intervention consists in 4 strength exercises: one will be performed into pain (ranging between 4 and 7 on NPRS scale) and the rest between 0 adn 2 on a NPRS scale
  Arms: exercising into pain
Other: exercising with no/slight pain — the intervention consists in 4 strength exercises and all of them will be performed in no pain/slight pain (between 0 and 2 on NPRS scale)
  Arms: exercising with no/slight pain

SUMMARY:
The aim of the randomized clinical trial is to investigate if "exercising into pain" gives better results in term of clinical outcomes compared to a non-painful exercise program.

DETAILED DESCRIPTION:
Exercise therapy is the first choice of treatment in the treatment of subacromial shoulder pain (SSP). Guidelines suggest exercise therapy for at least three months and research underlines the importance of progressive loaded exercise therapy at high dosage. However, it is not clear which is the best type of exercise and if pain should be provoked or avoided during exercise. Recent research found that painful exercises are beneficial in short term on pain and function in patients with different kinds of chronic musculoskeletal pain. The aim is to investigate if one painful exercise can give better and faster results in the management of SSP than non-painful program.

ELIGIBILITY:
Inclusion Criteria:

* shoulder pain for at least 3 months, elicited in the anterolateral shoulder region
* at least 3 out of 5 of the following tests positive: Neer test, Hawkins-Kennedy, Jobe, painful arc, external resistance test
* resting pain should be at 2/10 maximum on verbal numerical pain rating scale (NPRS)

Exclusion Criteria:

* bilateral shoulder pain
* corticosteroid injections 6 weeks prior to the study
* pregnancy, inability to understand spoken or written Dutch
* clinical signs of full-thickness rotator cuff tears (positive external and internal rotation lag tests and drop arm test)
* evidence of adhesive capsulitis
* previous cervical, thoracic or shoulder surgery; recent fractures or dislocations on the painful shoulder
* primary complaint of spinal pain or signs of central nervous system involvement or signs of cervical nerve root involvement; reproduction of shoulder pain with cervical rotation or axial compression
* primary diagnosis of acromioclavicular pathology, shoulder instability
* a radiologically confirmed fracture or previous medical imaging confirming the presence of calcification larger than 5 mm
* presence of competing pathologies (inflammatory arthritis, neurological disorders, fibromyalgia, malignancy, psychiatric illness, osteoporosis, hemophilia, rheumatic polymyalgia)
* more than 4h of training in sport overhead shoulder activities per week

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Change from baseline to 12 weeks
  There are 13 items, divided in two subscales: pain (5 items) and function (8 items). Each item is scored from 0 (no pain/no difficulty) to 10 (worst imaginable pain/so difficult it requires help) on a NPRS. The final score is a percentage derived from an average of the two subscales, where higher score means worse outcome.

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Change from baseline to 6 months
  There are 13 items, divided in two subscales: pain (5 items) and function (8 items). Each item is scored from 0 (no pain/no difficulty) to 10 (worst imaginable pain/so difficult it requires help) on a NPRS. The final score is a percentage derived from an average of the two subscales, where higher score means worse outcome.
Visual Analogue Scale (VAS) | Change from baseline to 12 weeks
  It measures pain during activity, during night, in the past 24 hours. It is measured on a scale from 0 to 100, where 0=no pain, 100=worst imaginable pain.
Visual Analogue Scale (VAS) | Change from baseline to 6 months
  It measures pain at rest, during activity, during night, in the past 24 hours. It is measured on a scale from 0 to 100, where 0=no pain, 100=worst imaginable pain.
Health-Related Quality of Life | Change from baseline to 12 weeks
  It is measured with: 1) EQ-5D-5L (EuroQol-5 dimentions-5 levels) index: score range from less than 0 (0=value of health state equivalent to dead; negative values indicate state worse than dead) to 1 (the value of full health), with higher scores indicating higher health; 2) EQ-5D VAS (EuroQol-5 dimentions-Visual Analogue Scale), from 0 to 100 score, with 0=lowest health-related quality of life, 100=best health-related quality of life)
Health-Related Quality of Life | Change from baseline to 6 months
  It is measured with: 1) EQ-5D-5L (EuroQol-5 dimentions-5 levels) index: score range from less than 0 (0=value of health state equivalent to dead; negative values indicate state worse than dead) to 1 (the value of full health), with higher scores indicating higher health; 2) EQ-5D VAS (EuroQol-5 dimentions-Visual Analogue Scale), from 0 to 100 score, with 0=lowest health-related quality of life, 100=best health-related quality of life)
Fear-Avoidance Beliefs Questionnaire (FABQ) | Change from baseline to 12 weeks
  It consists of 16 items and it has 2 subscales: Physical Activity (FABQ-PA, range: 0-24) and Work (FABQ-W, range: 0-42) higher scores mean more fear avoidance beliefs affecting physical activity and/or work.
Fear-Avoidance Beliefs Questionnaire (FABQ) | Change from baseline to 6 months
  It consists of 16 items and it has 2 subscales: Physical Activity (FABQ-PA, range: 0-24) and Work (FABQ-W, range: 0-42) higher scores mean more fear avoidance beliefs affecting physical activity and/or work.
Fear of Pain Questionnaire (FPQ-9) | Change from baseline to 12 weeks
  It is a shortened version of the Fear of Pain Questionnaire-III. The total score ranges between 9 and 45; higher scores mean more fear and anxiety associated with pain.
Fear of Pain Questionnaire (FPQ-9) | Change from baseline to 6 months
  It is a shortened version of the Fear of Pain Questionnaire-III. The total score ranges between 9 and 45; higher scores mean more fear and anxiety associated with pain.
Range of Movement (ROM) in internal rotation, external rotation, scaption | Change from baseline to 12 weeks
  It is measured with the inclinometer. The unit of measure is degrees.
Range of Movement (ROM) in internal rotation, external rotation, scaption | Change from baseline to 6 months
  It is measured with the inclinometer. The unit of measure is degrees.
Maximum Voluntary Contraction (MVC) in internal rotation, external rotation, scaption | Change from baseline to 12 weeks
  It is measured with the Hand-Held Dynamometer. The unit of measure is Newtons.
Maximum Voluntary Contraction (MVC) in internal rotation, external rotation, scaption | Change from baseline to 6 months
  It is measured with the Hand-Held Dynamometer. The unit of measure is Newtons.
Scapular Dyskinesis | Change from baseline to 12 weeks
  It is measured with visual observation at rest and during movement (loaded and unloaded, in abduction and in flexion); the presence of winging, tilting or abnormal scapular movement determines the judgement about scapular dyskinesis (yes/no) at rest and during movement
Scapular Dyskinesis | Change from baseline to 6 months
  It is measured with visual observation at rest and during movement (loaded and unloaded, in abduction and in flexion); the presence of winging, tilting or abnormal scapular movement determines the judgement about scapular dyskinesis (yes/no) at rest and during movement
Scapular Correction | Change from baseline to 12 weeks
  it is measured with the reduction of symptoms during 2 tests: 2) the scapular assistance test (SAT); if the pain reduces after the SAT, the test is considered positive; 3) scapular retraction test (SRT); if the pain reduces after the SRT, the test is considered positive.
Scapular Correction | Change from baseline to 6 months
  it is measured with the reduction of symptoms during 2 tests: 2) the scapular assistance test (SAT); if the pain reduces after the SAT, the test is considered positive; 3) scapular retraction test (SRT); if the pain reduces after the SRT, the test is considered positive.
Acromiohumeral Distance | Change from baseline to 12 weeks
  it is measured with the Ultrasound at 0 and 60 degrees of elevation in the scapular plane (in millimeters)
Acromiohumeral Distance | Change from baseline to 6 months
  it is measured with the Ultrasound at 0 and 60 degrees of elevation in the scapular plane (in millimeters)
Coracohumeral distance | Change from baseline to 12 weeks
  it is measured with the Ultrasound at 0 and 60 degrees of elevation in the scapular plane (in millimeters)
Coracohumeral distance | Change from baseline to 6 months
  it is measured with the Ultrasound at 0 and 60 degrees of elevation in the scapular plane (in millimeters)
Supraspinatus Tendon Thickness | Change from baseline to 12 weeks
  it is measured with the Ultrasound in Crass position (in millimeters)
Supraspinatus Tendon Thickness | Change from baseline to 6 months
  it is measured with the Ultrasound in Crass position (in millimeters)
Subscapularis Tendon Thickness | Change from baseline to 12 weeks
  it is measured with the Ultrasound in maximal external rotation (in millimeters)
Subscapularis Tendon Thickness | Change from baseline to 6 months
  it is measured with the Ultrasound in maximal external rotation (in millimeters)

OTHER OUTCOMES:
Global perceived effect (GPE) | 12 weeks
  It is measured on a 7-Likert Scale, ranging from 1 (way much better) to 7 (way much worse); higher scores mean worst global perceived effect.
Adherence | 12 weeks
  It is analysed in terms of attendance to the physiotherapist-led sessions and adherence to the home-exercise protocol. Good level of adherence is defined by: attendance of 7/9 (80%) of physiotherapist led-sessions and 22/27 (80%) days of home-exercises completed.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Struyf, Professor, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Physiotherapy private practices, Antwerp, Belgium

REFERENCES:
- [Derived] Cavaggion C, Navarro-Ledesma S, Juul-Kristensen B, Luque-Suarez A, Voogt L, Struyf F. The effect of painful exercise on ultrasonographic outcomes in rotator cuff-related shoulder pain: Secondary analysis of a randomized controlled trial. J Back Musculoskelet Rehabil. 2025 Nov;38(6):1379-1388. doi: 10.1177/10538127251334430. Epub 2025 May 14. PMID 40368129
- [Derived] Cavaggion C, Luque-Suarez A, Voogt L, Juul-Kristensen B, Wollants G, Beke L, Fransen E, Struyf F. Exercise into Pain in Chronic Rotator Cuff-Related Shoulder Pain: A Randomized Controlled Trial with 6-Month Follow-Up. Open Access J Sports Med. 2024 Nov 30;15:181-196. doi: 10.2147/OAJSM.S483272. eCollection 2024. PMID 39635498